CLINICAL TRIAL: NCT01777126
Title: A Simple Oral Nutrition Protocol Reduces Length of Stay in Patients With Regular Radical Cystectomy
Brief Title: Oral Nutrition After Regular Radical Cystectomy
Acronym: ONP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ONP
Record Dates: First submitted 2013-01-15; First posted 2013-01-28 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2011-01

CONDITIONS: Post Cystostomy
Keywords: cystectomy; parenteral nutrition; discharge; outcome
MeSH Terms: conditions — Hyperphagia | interventions — Population Groups; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Subjects enrolled in this arm will undergo usual medical and pharmaceutical care. In this group, parenteral nutrition (Oliclinomel N7) is part of the routine postoperative care program.
  Interventions: Other: Control group
- Oral Nutrition Protocol (ONP) group (Experimental): Oral intake was increased progressively with oral fluids and easily digestible food, independent of bowel movements. The corresponding energy content from the meals and oral fluids were calculated. Fortimel Jucy®, 200 ml containing 300 kcal, was used as the formulary energy sip. Extra fluids, up to two liter per day, were given intravenously, at the discretion of the treating physician. If the patient tolerated the ONP well, the oral intake was considered equal in terms of calories as the corresponding oral meal in the ONP. From the sixth day, the patient was allowed to eat at will. Only if oral intake remained insufficient after 5 days, which was left to the opinion of the treating physician, PN could be initiated in this group.
  Interventions: Other: Oral Nutrition Protocol (ONP) group

INTERVENTIONS:
Other: Oral Nutrition Protocol (ONP) group — For the experimental group, an oral nutrition protocol (ONP) with restrictive instructions for parenteral nutrition is implemented. Oral intake is increased progressively with oral fluids and easily digestible food, independent of clinical bowel movements. The oral energy sips used are Fortimel Jucy® (Nutricia) 200 ml containing 300 kcal. This provides supplementary energy and essential nutrients. Supplementary fluid, approximately up to two liter, is given intravenously. Only if oral intake is still insufficient after five days, PN (Oliclinomel N7) can be initiated.
  Arms: Oral Nutrition Protocol (ONP) group
Other: Control group — Subjects enrolled in this arm will undergo usual medical and pharmaceutical care. In this group, parenteral nutrition (Oliclinomel N7) is part of the routine postoperative care program.
  Arms: Control group

SUMMARY:
After radical cystectomy, postoperative ileus (POI) is a common complication resulting in a delayed oral nutritional intake with prolonged recovery and hospital stay. However, it is questionable if nutritional support by routine use of parenteral nutrition (PN) is justifiable.

A non-randomized before-after trial was conducted. Patients treated with an elective regular radical cystectomy and without preoperative contra-indications for enteral nutrition were eligible. In the control group, PN was initiated immediately after the procedure and continued until resumption of diet. In the interventional group, an ONP was implemented. PN could be initiated if oral intake was still insufficient after five days. The primary end point was the postoperative length of stay.

DETAILED DESCRIPTION:
Design

A prospective interventional non-randomized before-after trial was conducted. Eligible patients admitted from 01/02/2009 were consecutively assigned to the control group until the predefined sample size was reached. After enrollment and follow-up of control patients had been finished, all newly admitted eligible patients were consecutively assigned to the interventional group.

In addition to the before-after study, a sample of eligible patients was collected from March 2011 to March 2013 (follow-up group) to examine the post-study impact of the ONP.

Patients

All adult patients admitted to the 48-bed urological ward in the 1850 bed University Hospitals Leuven and treated with elective and regular RC, whether or not for underlying cancer, were eligible for inclusion. Three different diversions are performed: an ileal conduit, an orthothopic neobladder (N-pouch)12 or a continent cutaneous diversion. The surgical procedure was considered regular if the patient returned after the procedure to the urological ward and was not transferred to the intensive care unit. If the latter was deemed necessary by the treating surgeon, the patient would be subjected to the intensive care nutrition protocol. Therefore, only regular RC patients were included.

Exclusion criteria were transfer to the intensive care unit, preoperative contra-indications for EN and discharge to a rehabilitation center. Contra-indications for EN were defined as intestinal obstruction, malabsorption, multiple high-output fistula or intestinal ischemia8. Uretero-ileal or ileo-ileal anastomoses, resulting from RC, were not considered as a contra-indication for EN9,10. Discharge to a rehabilitation center could surpass one of the criteria for discharge, i.e. the ability of independent mobilization, and could therefore influence the postoperative LOS.

Care practices other than nutrition management

Preoperatively, all patients received bowel preparation with a 2 liter osmotic laxative (macrogol 3350 100 g, sodiumsulphate 7.5 g, NaCl 2.69 g, KCl 1.02 g, sodium salt of ascorbic acid 5.9 g and ascorbic acid 4.7 g). Before incision, a loading dose of 0.05 ml/cm epidural analgesics (levobupivacaine 2,5 mg/ml and sufentanil 1 mcg/ml) was administered. During surgery, a central venous catheter, a nasogastric or percutaneous gastrostomy tube and ureteral stents were inserted. The nasogastric or percutaneous gastrostomy tube was removed on the first or second postoperative day after restoration of transit (defined as a residual gastric volume of less than 50 ml/24h). Acetaminophen, non-steroidal anti-inflammatory drugs and patient-controlled epidural analgesia (PCEA; levobupivacaine 2,5 mg/ml and sufentanil 1 mcg/ml) were available for postoperative acute pain management. Intraoperative antimicrobial prophylaxis consisted of cefazoline and metronidazole. Thromboprophylaxis consisted of enoxaparin. Anti-emetics and other prokinetic drugs were not routinely administered but only prescribed when needed. All treating surgeons were fully trained at the start of the study.

After a minimum of 10 days, ureteral stents were removed if the following 3 criteria were met: restoration of transit, presence of bowel movements and absence of fever (defined as body temperature <38,3 °C). Prophylactic levofloxacin 500 mg once daily was administered after stent removal, until the first consultation. Patients were discharged if the following 4 criteria were fulfilled: 1) removal of all drains and stents, 2) the absence of fever (body temperature < 38,3 °C), 3) the ability to tolerate solid food and 4) the ability of independent mobilization.

The abovementioned care practices (anesthesia modalities, surgical techniques, doses of narcotics, bowel stimulants and anti-nauseants, and mobilization practices) did not alter during the course of the study.

Nutrition management

In the control group, PN was initiated immediately after surgery and continued until the patient was able to tolerate solid food. PN infusion therapy consisted of Olimel® (Baxter S.A., Lessines, Belgium) N7E 1000 ml, 1500 ml or 2000 ml; a parenteral solution with a total energy of 1100 kcal/1000 ml and containing polyamino-acids (43.75g/1000 ml), glucose (140g/1000ml), lipids (40g/1000ml) and electrolytes. Cernevit® (Baxter S.A., Lessines, Belgium), a multivitamin powder for injection, and Addamel® (Fresenius Kabi, Schelle, Belgium), a concentrate for injection containing trace elements, were added daily to the PN. The amount of PN administered depended on the non-protein requirements, calculated by 30 ± 10% kcal/kg ideal body weight13. Extra fluids, up to two liter per day, were given intravenously, at the discretion of the treating physician.

In the interventional group, the ONP was implemented (Table 1). Oral intake was increased progressively with oral fluids and easily digestible food, independent of bowel movements. The corresponding energy content from the meals and oral fluids were calculated. Fortimel Jucy®, 200 ml containing 300 kcal, was used as the formulary energy sip. Extra fluids, up to two liter per day, were given intravenously, at the discretion of the treating physician. Nurses verified daily whether the patient was able to tolerate the ONP. If the patient tolerated the ONP well, the oral intake was considered equal in terms of calories as the corresponding oral meal in the ONP. From the sixth day, the patient was allowed to eat at will. Only if oral intake remained insufficient after 5 days, which was left to the opinion of the treating physician, PN could be initiated in this group.

Data collection

The following baseline demographic data were retrieved from medical files: patient characteristics (gender, age, weight, length, body mass index, age-adjusted Charlson comorbidity index14, indication for RC (oncologic or neurogenic) and bladder cancer staging (TNM classification15)), surgical aspects (type of urinary diversion, attending surgeon, intra-operative blood loss and duration of procedure), postoperative ileus (POI) and day of nasogastric tube removal. The age-adjusted Charlson comorbidity index is a method for classifying comorbid conditions. As the increase in elderly population and concurrent increase in oncologic disease (and thus in bladder cancer) emphasized the importance of understanding the interaction between age an comorbid illness on life expectancy, the age -adjusted version was used. POI was defined as the inability to tolerate solid food, the need to place a nasogastric tube in suction, the need to stop oral intake due to abdominal distention (evaluated by the treating clinician), nausea or emesis.

Endpoints

The primary endpoint was LOS from surgery to discharge.

Secondary endpoints were the number of patients with successful implementation of the ONP, as well as number of administered PN infusion bags per patient, time to resumption of full diet, number of patients with one or more postoperative complications (POC), number of POCs per patient, type and severity grade of POCs and the incidence of catheter related bloodstream infections (CRBSIs). The implementation of the ONP was considered successful if the protocol could be completely applied and no PN was needed. The type and severity of POCs were classified using the Clavien-Dindo classification16. POCs were classified into 11 categories and stratified by severity. CRBSI, a common PN-related complication6, was defined as bacteremia or fungemia in a patient having an intravascular device and more than one positive blood culture result obtained from a peripheral vein, clinical manifestations of infection (e.g., fever, chills, and/or hypotension) and no apparent other source for blood stream infection17.

Post-study impact

An additional patient cohort was assembled, using the same inclusion and exclusion criteria as described above. The LOS and number of PN infusion bags after surgery were determined and compared to the results obtained from the intervention group.

Analysis of PN associated costs

The avoided PN cost per patient were calculated. For every group, the total number of PN infusion bags was divided by the number of patients and multiplied by € 60, which was the average actual cost in euros of one bag of Olimel® in Belgium at the time of the study. This resulted in a direct and comparable PN infusion bag related cost per patient per group.

Statistical analysis and sample size calculation

Statistical analysis was performed by L-Biostat, Catholic University Leuven, using SPSS package (SPSS Statistics 20.0 for Windows). Chi-square and Fisher's Exact tests were used for categorical data. The unpaired T-test or the Wilcoxon rank sum test was used for normal and non-normal distributed continuous variables respectively. Baseline demographic data and the outcome measures were considered statistically significant if p-values were < 0.05. The Bonferroni correction was used to account for multiple comparisons (6 secondary outcome measures). Therefore, secondary outcome parameters were considered statistically significant if p-values were < 0.008. To asses factors influencing LOS, general linear model statistics - univariate analysis followed by ANOVA - were carried out.

Preliminary data from our institution showed that all RC patients receiving PN directly after surgery were discharged after a mean of 19.3 ± 5.6 days. We expected to reduce our LOS with 3 days from 19 to 16 days by implementing the ONP. Assuming that variances for both groups are comparable, 88 (2x44) patients were needed, giving at least 80 % power (α=0.05, one-tailed) to reject the null hypothesis defined as no difference in postoperative LOS between the two groups.

The study was approved by the hospital's Ethics Committee and registered on clinical trials.gov n° NCT01777126. No informed consent was obtained as the introduction of the ONP was part of continuous improvement of standard of care in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* regular radical cystectomy

Exclusion Criteria:

* preoperative contra-indications for enteral nutrition (EN): intestinal obstruction, malabsorption, multiple high-output fistula and intestinal ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Declercq, Pharm.D, Principal Investigator — Pharmacy Department, University Hospitals Leuven & Department of Pharmaceutical and Pharmacological Sciences, KULeuven, Belgium
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult patients admitted undergoing an elective and unproblematic radical cystectomystarting in 01/02/2009 were consecutively assigned to the control group until the predefined sample size was attained. After completion of the control group, all newly admitted patients were, again consecutively, assigned to the experimental group.
Pre-assignment Details: If a transfer was needed, the patient was excluded. Other exclusion criteria were preoperative contra-indications for EN and discharge to a rehabilitation center.
Groups:
- Control Group: In the control group, PN was part of the routine postoperative care pathway. PN was initiated the day postoperatively and was continued until the patients were able to tolerate solid food. PN consisted of Olimel® N7E 1000, 1500 ml or 2000 ml, a parenteral solution with a non-protein energy of 960 kcal/1000ml and containing polyamino-acids (43.75g/1000 ml), glucose (140g/1000ml), lipids (40g/1000ml) and electrolytes. The amount of PN administered depended on non-protein requirement, calculated by 25 kcal/kg ideal body weight ± 10%. Cernevit®, a multivitamin powder for injection, and Addamel®, a trace elements containing concentrate for injection, were added to the PN daily. Supplementary fluids, up to two liter per day, was given intravenously, if deemed necessary by the treating physician.
- Oral Nutrition Protocol (ONP) Group: In this group, oral intake was increased progressively with oral fluids and easily digestible food, independent of clinical bowel movements. The oral energy sips used were Fortimel Juicy®, 200 ml containing 300 kcal (total energy). A detailed description of the content of Fortimel Jucy® is available on www.nutriciamedical.be. Supplementary fluids, up to two liter per day, was given intravenously, if deemed necessary by the treating physician. If the patient was unable to produce stools on the third day post-surgery, neostigmine (Prostigmine® 0.5 mg subcutaneous, maximum four times a day), promoting the movement of intestinal contents by augmenting motor activity of the small and large bowel [14], could be administered. Only if oral intake was still insufficient after five days, as defined by the opinion of the treating physician, PN could be initiated in this group.
Period: Overall Study
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Started | 48 | 46
Completed | 48 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Subjects enrolled in this arm will undergo the routine postoperative care pathway. PN was initiated the day postoperatively and was continued until the patients were able to tolerate solid food. PN consisted of Olimel® N7E 1000, 1500 ml or 2000 ml, a parenteral solution with a non-protein energy of 960 kcal/1000ml and containing polyamino-acids (43.75g/1000 ml), glucose (140g/1000ml), lipids (40g/1000ml) and electrolytes. The amount of PN administered depended on non-protein requirement, calculated by 25 kcal/kg ideal body weight ± 10%. Cernevit®, a multivitamin powder for injection, and Addamel®, a trace elements containing concentrate for injection, were added to the PN daily. Supplementary fluids, up to two liter per day, was given intravenously, if deemed necessary by the treating physician.
- Oral Nutrition Protocol (ONP) Group: Subjects enrolled in this arm will undergo the ONP protocol. Oral intake was increased progressively with oral fluids and easily digestible food, independent of clinical bowel movements. The oral energy sips used were Fortimel Juicy®, 200 ml containing 300 kcal (total energy). A detailed description of the content of Fortimel Jucy® is available on www.nutriciamedical.be. Supplementary fluids, up to two liter per day, was given intravenously, if deemed necessary by the treating physician. If the patient was unable to produce stools on the third day post-surgery, neostigmine (Prostigmine® 0.5 mg subcutaneous, maximum four times a day), promoting the movement of intestinal contents by augmenting motor activity of the small and large bowel [14], could be administered. Only if oral intake was still insufficient after five days, as defined by the opinion of the treating physician, PN could be initiated in this group.
- Total: Total of all reporting groups
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 66.0 (12.5) [55 to 75] | 65.5 (10.8) [57 to 72.5] | 66 (11.6) [55.75 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 31 | 34 | 65
Length [Mean (Standard Deviation); unit: cm] | 169.7 (8.2) | 170.8 (8.0) | 170.3 (8.1)
Weight [Mean (Standard Deviation); unit: kg] | 73.7 (13.9) | 75.4 (14.2) | 74.6 (14.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 25.5 (4.0) | 25.8 (4.3) | 25.7 (4.1)
Age-adjusted Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: Points] — The Age-adjusted Charlson Comorbidity index encompasses 19 medical conditions weighted 1-6 with total scores ranging from 0-37. Mortality for each disease was converted to a relative risk of death within 12 months and a weight was then assigned. From the weighted conditions, a sum score can be tallied to yield the total comorbidity score. The CCI can be further adapted to account for increasing age. To account for the effects of increasing age, one point can be added to the CCI score for each decade of life over the age of 50 [13].
  Points | 4 (1.7) [3 to 5] | 5 (2.6) [3 to 6] | 4 (2.3) [3 to 6]
Indication [Number; unit: participants]
  Neurogenic | 9 | 6 | 15
  Oncologic | 39 | 40 | 79
Bladder staging [Number; unit: participants] — The TNM system has been widely adopted in bladder staging. The number of Ts Ns and Ms depend on the tumour / site.
  T: Tumour N: Node M: Metastases
  participants
    T+N0M0 | 1 | 1 | 2
    T+N+M0 | 1 | 0 | 1
    T+N+M+ | 38 | 40 | 78
    T0N0M0 | 8 | 5 | 13
Type of urinary diversion [Number; unit: participants]
  Ileal conduit | 40 | 39 | 79
  Orthothopic neobladder | 6 | 7 | 13
  Continent cutaneous diversion | 2 | 0 | 2
Surgeon [Number; unit: participants]
  Surgeon 1. | 5 | 0 | 5
  Surgeon 2. | 19 | 14 | 33
  Surgeon 3. | 5 | 3 | 8
  Surgeon 4. | 19 | 29 | 48
Blood loss [Median (Inter-Quartile Range); unit: ml] — Volume of blood loss during surgery.
  ml | 1000 (600) [500 to 1475] | 1000 (589) [600 to 1650] | 1000 (595) [575 to 1500]
Duration of procedure [Median (Inter-Quartile Range); unit: minute] | 210 (55.4) [180 to 240] | 187.5 (46.8) [180 to 240] | 210 (51.1) [180 to 240]
Postoperative ileus [Number; unit: participants] — Postoperative ileus was defined as the inability to tolerate solid food, the need to place a nasogastric tube in suction or the need to stop oral intake due to abdominal distention, nausea or emesis.
  participants
    POI | 9 | 13 | 22
    no POI | 39 | 33 | 72
Nasogastric tube removal day [Median (Inter-Quartile Range); unit: day] | 2 [1 to 4.75] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: the Postoperative Length of Stay
Description: The primary outcome measure was the interval from surgery to discharge. Discharge means that the patient returns to his home.
Time Frame: one month after surgery
Population: Primary outcome measure was interval from surgery to discharge. Discharge means that the patient returns back to his home and not to a rehabilitation center.
Measure: Median (Inter-Quartile Range); unit: day
Groups:
- Control Group: For subjects enrolled in this arm, PN was part of the routine postoperative care pathway. PN was initiated the day postoperatively and was continued until the patients were able to tolerate solid food. PN consisted of Olimel® N7E 1000, 1500 ml or 2000 ml, a parenteral solution with a non-protein energy of 960 kcal/1000ml and containing polyamino-acids (43.75g/1000 ml), glucose (140g/1000ml), lipids (40g/1000ml) and electrolytes. The amount of PN administered depended on non-protein requirement, calculated by 25 kcal/kg ideal body weight ± 10%. Cernevit®, a multivitamin powder for injection, and Addamel®, a trace elements containing concentrate for injection, were added to the PN daily. Supplementary fluids, up to two liter per day, was given intravenously, if deemed necessary by the treating physician.
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
day | 18 (5.6) [15 to 22] | 14 (4.3) [13 to 18]
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; The primary outcome measure was the interval from surgery to discharge. Discharge means that the patient returns to his home. Preliminary data from our institution showed that all patients received parenteral nutrition very early post-surgery and were discharged after a mean of 19.3 ± 5.6 days. Therefore, the primary objective by implementing the ONP was to reduce the length of stay with 3 days; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 3

2. Secondary Outcome: Successful Implementation Rate of the ONP in the Experimental Group
Description: Successful implementation of the ONP was achieved if the patient followed the protocol and did not need PN.
Time Frame: 30 days postoperative
Population: The number of patients with successful implementation of the ONP in the experimental group.
Measure: Number; unit: participants
Arm/Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 46
participants | 40

3. Secondary Outcome: Number of Administered PN
Description: Number of administered PN per group
Time Frame: 30 days postoperative
Measure: Number; unit: number of PN
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
number of PN | 435 | 24

4. Secondary Outcome: The Time to Resumption of Full Diet.
Description: The time to resumption of full diet between the two groups was compared.
Time Frame: 30 days postoperative
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
day | 8 [6 to 9] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; Statistical analysis was performed by the Leuven Statistics Research Centre, KU Leuven, using SPSS package (SPSS Statistics 20.0 for Windows). Statistical analysis was performed using the Wilcoxon rank sum test. The result was considered statistically significant if p-values were < 0.05; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4

5. Secondary Outcome: Patients With One or More Postoperative Complication.
Description: Number of patients with one or more postoperative complication were compared betweent the two groups.
Time Frame: 30 days postoperative
Measure: Number; unit: participants
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
participants | 37 | 32
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; Statistical analysis was performed by the Leuven Statistics Research Centre, KU Leuven, using SPSS package (SPSS Statistics 20.0 for Windows). Statistical analysis was performed using Chi-square and Fisher's Exact Test. Results were considered statistically significant if p-values were < 0.05; Test type: Superiority or Other; p = 0.487, Fisher Exact; proportion

6. Secondary Outcome: The Number of Postoperative Complications Per Patient.
Description: The number of postoperative complications per patient was compared between the two groups.
Time Frame: 30 days postoperative
Measure: Median (Inter-Quartile Range); unit: number of postoperative complications
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
number of postoperative complications | 1 [1 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; Test type: Superiority or Other; p = 0.302, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0

7. Secondary Outcome: Patients With a Catheter Related Bloodstream Infection
Description: Patients with a catheter related bloodstream infection were compared between the two groups
Time Frame: 30 days postoperative
Measure: Number; unit: participants
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
participants | 4 | 0
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; Statistical analysis was performed by the Leuven Statistics Research Centre, KU Leuven, using SPSS package (SPSS Statistics 20.0 for Windows). Statistical analysis was performed using Fisher's Exact Test. The result was considered statistically significant if p-values were < 0.05; Test type: Superiority or Other; p = 0.117, Fisher Exact; Proportion

8. Secondary Outcome: The Type of Postoperative Complications.
Description: The type of postoperative complications (POCs) were compared between the two groups. The type of POCs were classified using the Clavien-Dindo Classification. Herein POCs were classified into 8 categories (1. Infection, 2. Fistula/leak, 3. Bleeding/hematoma, 4. Gastrointestinal, 5. Cardiopulmonary, 6. Neurologic, 7. pain and 8. Other) and stratified by their severity grade (Table 2). Per patient, multiple complications are possible.
Time Frame: 30 days postoperative
Measure: Number; unit: number per type of POC
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
number per type of POC
  1. Infection | 21 | 13
  2. Fistula or leak | 1 | 2
  3. Bleeding or hematoma | 5 | 2
  4. Gastro-intestinal | 13 | 16
  5. Cardiopulmonary | 13 | 4
  6. Neurologic | 0 | 5
  7. Pain | 2 | 0
  8. Other | 15 | 11
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; Statistical analysis was performed by the Leuven Statistics Research Centre, KU Leuven, using SPSS package (SPSS Statistics 20.0 for Windows). Statistical analysis was performed using Chi-square Test. Outcome measures were considered statistically significant if p-values were < 0.05; Test type: Superiority or Other; p = 0.049, Chi-squared; Proportion

9. Secondary Outcome: Severity Grade of Postoperative Complications.
Description: Severity grade of postoperative complications (POCs) was compared between the two groups. The severity grade of POCs were classified using the Clavien-Dindo Classification. Per patient, multiple complications are possible.
Time Frame: 30 days postoperative
Measure: Number; unit: number of POCs per severity grade
Arm/Group | Control Group | Oral Nutrition Protocol (ONP) Group
Number analyzed (Participants) | 48 | 46
number of POCs per severity grade
  Severity Grade 1 Clavien Dindo | 15 | 16
  Severity Grade 2 Clavin Dindo | 35 | 23
  Severity Grade 3a Clavien Dindo | 16 | 12
  Severtity Grade 3b Clavine Dindo | 4 | 2
Statistical Analysis 1: Comparison: Control Group vs Oral Nutrition Protocol (ONP) Group; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.698, Chi-squared; proportion

ADVERSE EVENTS:
Time Frame: 30 days
Description: Number of patients with one or more postoperative complications (POC), number of POCs per patient and type and severity grade of POCs.
  The type and severity of POCs were classified using the Clavien-Dindo classification16. POCs were classified into 11 categories and stratified by severity.
Groups:
- Enhanced Recovery Oral Nutrition Protocol (ERONP) Group: Subjects enrolled in this arm will undergo the ERONP protocol. An enhanced oral nutrition protocol (ERONP) with restrictive instructions for parenteral nutrition is implemented. Oral intake is increased progressively with oral fluids and easily digestible food, independent of clinical bowel movements. The oral energy sips used are Fortimel Juicy® (Nutricia) 200 ml containing 300 kcal. This provides supplementary energy and essential nutrients. Supplementary fluid, approximately up to two liter, is given intravenously. If the patient is unable to produce stools on the third day post-surgery, neostigmine (Prostigmin® 0.5 mg subcutaneous, maximum 4 times a day), an acetylcholinesterase inhibitor promoting the movement of intestinal contents by augmenting motor activity of the small and large bowel, can be administered. Only if oral intake is still insufficient after five days, PN (Oliclinomel N7) can be initiated.
Arm/Group | Control Group | Enhanced Recovery Oral Nutrition Protocol (ERONP) Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 37/48 | 32/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=48) | Enhanced Recovery Oral Nutrition Protocol (ERONP) Group (N=46)
Infection (Infections and infestations) | 20 (21) | 13 (13)
Fistula or leak (General disorders) | 1 (1) | 2 (2)
Bleeding (General disorders) | 5 (5) | 2 (2)
DGE/Nausea&vomiting (Gastrointestinal disorders) | 10 (13) | 15 (16)
Cardiopulmonary (Cardiac disorders) | 11 (12) | 4 (4)
Neurologic (Nervous system disorders) | 0 (0) | 3 (5)
Pain (General disorders) | 2 (2) | 0 (0)
Other (General disorders) | 13 (15) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes